CLINICAL TRIAL: NCT04349657
Title: An RCT Evaluating the Safety and Efficacy of the Endovascular Treatment of Subjects with Stenotic or Restenotic Lesions of the Common Femoral Artery with the Supera Vascular Mimetic Implant Compared to Surgical Common Femoral Artery Endarterectomy
Brief Title: A Study Evaluating the Endovascular Treatment of Subjects with Stenotic or Restenotic Lesions of the Common Femoral Artery with the Supera Vascular Mimetic Implant Compared to Surgical Common Femoral Artery Endarterectomy
Acronym: SUPERSURG-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPERSURG RCT-v1.0-05MAR2020
Record Dates: First submitted 2020-04-09; First posted 2020-04-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly assigned in a 1:1 manner to treatment with either the Supera stent or endarterectomy.
Masking Description: All parties will know in what arm the study subject is randomized before the study procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supera Peripheral Stent System treatment group (Experimental): These patients will be treated endovascularly with the Supera Peripheral Stent System (Abbott).
  Interventions: Device: Supera Peripheral Stent System treatment group
- Endarterectomy treatment group (Active Comparator): These patients will be treated surgically with endarterectomy
  Interventions: Procedure: Endarterectomy treatment group

INTERVENTIONS:
Device: Supera Peripheral Stent System treatment group — Percutaneous endovascular stenting with the Supera Peripheral Stent System
  Arms: Supera Peripheral Stent System treatment group
Procedure: Endarterectomy treatment group — Surgical treatment through endarterectomy
  Arms: Endarterectomy treatment group

SUMMARY:
The SUPERSURG RCT trial investigates the efficacy and safety of the endovascular treatment of stenosis or restenosis in the common femoral artery (CFA) of patients presenting with Rutherford classification 2,3 or 4 with a Supera Vascular Mimetic Implant of Abbott, compared to classic surgical common femoral artery endarterectomy. The Supera Vascular Mimetic Implant has an interwoven design and has a high crush resistance and is, when correctly implanted, an ideal stent to treat eccentric calcified plaques in the CFA.

An expected total of 143 patients will be treated with the Vascular Mimetic Implant of Abbott and compared to a control group of another 143 patients that will be treated with classic surgical endarterectomy of the common femoral artery. Assignment to the treatment groups will be at random.

Patients will be invited for a follow-up visit at 1, 6, 12, 24 and 36 months post-procedure.

The primary efficacy endpoint is defined as follows: freedom from clinically-driven target lesion revascularization and binary restenosis at 12 months. The primary safety endpoint is defined as follows: a composite of overall death, cardiac, pulmonary, renal complications, sepsis, target lesion revascularisation and wound related complications through 30 days post-index procedure.

The secondary endpoints are defined as technical success, primary patency in the deep femoral artery, primary patency in the target lesion, target lesion revascularisation, target vessel revascularisation, binary restenosis, duration of initial hospital stay, sustained clinical improvement, change of walking impairment questionnaire score from baseline, change in target limb Rutherford classification, change in target limb ABI/TBI from baseline, all cause death, thrombosis at the target lesion through 6, 12, 24 and 36 months post-procedure.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to assess the safety and efficacy of the Supera Vascular Mimetic Implant for the treatment of stenotic or restenotic lesions of the common femoral artery. Furthermore, a non-inferiority hypothesis in terms of efficacy and a superiority in terms of safety will be tested with the endovascular treatment with Supera compared to surgical endarterectomy of the common femoral artery.

The patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should be geographically stable, willing and able to cooperate in this clinical study, and remain available for long term follow-up. The patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful guidewire passage through the study target lesion.

Prior to the index procedure the following will be collected: an informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of acute limb ischemia (Rutherford category), the resting ankle-brachial index (ABI) or toe-brachial index (TBI), blood sample test (complete blood count, comprehensive metabolic panel and if applicable pregnancy test) and a walking impairment questionnaire. Randomization will also occur prior to the procedure.

During the procedure patients that are randomized within the endarterectomy group will be treated according to the institutions standard of care. For patients that are randomized within the Supera arm, the guidewire will cross the entire study lesion after which the lesion will be assessed through angiography. Pre-dilatation of the target lesion with an uncoated PTA-balloon is mandatory and will be followed by stenting with the Supera stent according to the instructions for use. Postdilatation of the stent is allowed but not mandatory.

The regular follow-up is necessary to monitor the condition of the patient and the results of the procedure. The patients will be invited for the following required follow-up visits at 1, 6, 12, 24 and 36 months. During these visit the following data will be collected: medication record, physical exam, target limb ABI/TBI and Rutherford classification, duplex ultrasound of target vessel, walking impairment questionnaire and possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years old
* Patient presenting a score from 2 to 4 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a life expectancy of at least 12 months
* Prior to enrolment, the guidewire has crossed the target lesion in the endovascular arm. In the surgical arm, the endarterectomy needs to be performed with primary suture or patch implantation
* De novo stenotic or restenotic (post-PTA) lesions (<100%) located in the common femoral artery, suitable for both endovascular therapy and endarterectomy
* Target lesion is located within the native CFA: localized between 1cm proximal to the origin of the circumflex iliac artery and the proximal (2cm) superficial femoral artery and deep femoral artery (2cm) (Azéma type 2 and 3 lesions)
* There is angiographic evidence of a patent deep femoral artery and/or superficial femoral artery
* The target lesion has angiographic evidence of >50% stenosis. Occlusions are not allowed.

Exclusion Criteria:

* Presence of another stent in the target vessel that was placed during a previous procedure
* Previous open surgery in the ipsilateral groin
* Patients contraindicated for antiplatelet therapy, anticoagulants or thrombolytics
* Patients who exhibit persistent acute intraluminal thrombus at the target lesion site
* Patients with known hypersensitivity to nickel-titanium and heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Known allergy to contrast media that cannot be adequately pre-medicated prior to study procedure
* Patients with uncorrected bleeding disorders
* Female patients with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Ipsilateral inflow (aorto-iliac) artery treatment before target lesion treatment with a residual stenosis >30%
* Use of thrombectomy, atherectomy or laser device during procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Severe medical comorbidities (untreated coronary artery disease/congestive heart failure, severe chronic obstructive pulmonary disease, metastatic malignancy, dementia, etc.) or other medical condition that would prelude compliance with the study protocol or 1-year life expectancy
* Major distal amputation (above the ankle) in the study limb or non-study limb
* Target lesion involves an (pseudo-)aneurysm or is adjacent to an (pseudo-)aneurysm (within 5mm)
* Iliac inflow disease requiring treatment, unless the iliac artery disease is successfully treated first during the index procedure. Success is defined as ≤30% residual diameter stenosis without death or major complications
* Presence of an aortic, iliac or femoral artificial graft
* Occlusion in the target lesion
* Presence of an interposition graft with/without profunda reimplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint at 12 months: Primary patency | 12 months post-index-procedure
  To demonstrate the non-inferior efficacy in the group treated with the Supera stent compared to the group treated with endarterectomy for the treatment of atherosclerosis in the common femoral artery (CFA). Efficacy is defined as primary patency: freedom from restenosis defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4 or ≥50% stenosis as assessed by an independent DUS core lab in CFA without a previous target lesion revascularization through 12 months post-index procedure.
Primary safety endpoint at 30 days post-index procedure | 30 days post-index-procedure
  To demonstrate superior safety in the group treated with the Supera stent compared to the endarterectomy group for the treatment of atherosclerosis in the CFA. Safety is defined as a composite of overall death, cardiac, pulmonary, renal complications, sepsis, target lesion revascularization (TLR) and wound-related complications (haematoma, seroma, lymphocele, lymphatic leaks with lymphatic fistula, surgical site infections (SSIs) (Szilagyi grade I, II and III)).

SECONDARY OUTCOMES:
Technical success: post-procedure residual stenosis <30% | Index procedure
  Supera group: Defined as the ability to cross and stent the lesion to achieve residual angiographic stenosis no greater than 30%.
  Endarterectomy group: defined as the ability to remove the atherosclerotic plaque with or without patch (interposition grafts are not allowed). In the imaging subcohort the endarterectomy is considered successful when a residual stenosis no greater than 30% per visual estimation is confirmed.
Primary patency in the deep femoral artery (DFA), post-index procedure and at 6-, 12-, 24- and 36-months post-index procedure | 6, 12, 24 and 36 months post-index-procedure
  Primary patency in the DFA is defined as freedom from an occlusion in the DFA as assessed by PSV-values. This PSV-value will be assessed pre-procedure, post-procedure, 6 months and 12 months post-index procedure. At 12 months, the PSV-value will be core-lab controlled.
Primary patency at 6, 24 and 36 months | 6, 24 and 36 months post-index-procedure
  Primary patency is a composite of freedom from clinically-driven target lesion revascularization (CD-TLR) and binary restenosis (restenosis defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4 or ≥50% stenosis as assessed by DUS in CFA) through 6 months post-index procedure
TLR at 6-, 12-, 24- and 36-months post-index procedure | 6, 12, 24 and 36 months post-index-procedure
  TLR is defined as a reintervention to maintain or restore the patency in the target lesion. TLR is clinically-driven (CD) when the TLR was needed due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure
TVR at 6-, 12-, 24- and 36-months post-index procedure | 6, 12, 24 and 36 months post-index-procedure
  Target vessel revascularization (TVR) is defined as a reintervention to maintain or restore the patency in the target vessel. TVR is clinically-driven (CD) when the TVR was needed due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure
Binary restenosis at 6, 12, 24 and 36 months | 6, 12, 24 and 36 months post-index-procedure
  Binary restenosis is defined as restenosis confirmed by DUS PSVR ≥2.4 or ≥50% stenosis as assessed by angiographic and DUS images. At 12 months, the images will be core lab controlled
Duration of initial hospitalisation stay | Up to 4 weeks
  Number of hours/days of the initial hospitalisation stay.
Sustained clinical improvement at 6-, 12-, 24- and 36-months post-index procedure | 6, 12, 24 and 36 months post-index-procedure
  Clinical improvement is defined as freedom from major target limb amputation, TVR, worsening target limb Rutherford class (compared to baseline) and decrease in target limb ankle brachial index (ABI) or toe brachial index (TBI) ≥0.15 (compared to baseline)
Change in Walking Impairment Questionnaire (WIQ) score from baseline to 6, 12, 24 and 36 months | 6, 12, 24 and 36 months post-index-procedure
  change in walking impairment questionnaire (WIQ) score from baseline to 6 and 12 months.
  The WIQ consists of 6 sections each consisting of multiple questions. Each question is scored from 0 to 4 (0 meaning a lot of problems and 4 no problems at all). The scores per section are summed up and recalculated to percentages (100% meaning very good and 0% meaning very bad). All the sections are averaged to give the final WIQ-score.
Change in target limb Rutherford class from baseline to 6, 12, 24 and 36 months | 6, 12, 24 and 36 months post-index-procedure
  Change in target limb Rutherford class from baseline to 6, 12, 24 and 36 months
Change in target limb resting ABI or TBI from baseline to 6, 12, 24 and 36 months | 6, 12, 24 and 36 months post-index-procedure
  Change in target limb resting ABI or TBI from baseline to 6, 12, 24 and 36 months
All cause death at 6, 12, 24 and 36 months | 6, 12, 24 and 36 months post-index-procedure
  All cause death at 6, 12, 24 and 36 months
Thrombosis at the target lesion at 6, 12, 24 and 36 months | 6, 12, 24 and 36 months post-index-procedure
  Thrombosis at the target lesion at 6, 12, 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — A.Z. Sint-Blasius
Locations (13):
- Belgium (7):
  - O.L.V. Hospital, Aalst
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
  - Z.O.L., Genk
  - Az Groeninge, Kortrijk
  - AZ Sint-Maarten, Mechelen
  - A.Z. Jan Portaels, Vilvoorde
- Netherlands (4):
  - Maastricht UMC+, Maastricht, Limburg
  - Dijklander hospital, Hoorn, North Holland
  - St Antonius Hospital, Utrecht, Utrecht
  - Noordwest ziekenhuisgroep, Alkmaar
- Poland (2):
  - Bonifraterskie Centrum Medyczne, Krakow
  - Karol Marcinkowski Medical University, Poznan

IPD SHARING:
Plan to Share IPD: No